CLINICAL TRIAL: NCT00005797
Title: Allogeneic Bone Marrow Transplantation for Hematologic Malignancies: A Treatment Approach Based on Risk of Relapse and Toxicity
Brief Title: Bone Marrow Transplant in Treating Patients With Hematologic Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-11281; MCC-IRB-4188 (Other: University of South Florida); NCI-G00-1759 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2012-10

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Multiple Myeloma and Malignant Plasma Cell Neoplasms; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: refractory multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; refractory chronic lymphocytic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; polycythemia vera; primary myelofibrosis; essential thrombocythemia; refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; previously treated myelodysplastic syndromes; refractory cytopenia with multilineage dysplasia; chronic eosinophilic leukemia; chronic neutrophilic leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Multiple Myeloma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Congenital Abnormalities | interventions — Busulfan; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BuCy2 (Other): Busulfan & Cyclophosphamide
  Interventions: Drug: busulfan; Drug: Cyclophosphamide
- VP16/TBI (Other): Fractionated Total Body Irradiation + VP-16
  Interventions: Drug: VP-16; Radiation: Fractionated Total Body Irradiation (FTBI)

INTERVENTIONS:
Drug: busulfan — administered on Day -7 through Day -4. The total dose is 12.8 mg/kg
  Other Names: Busulfex®
  Arms: BuCy2
Drug: Cyclophosphamide — administered at a dose of 60 mg/kg on each of two successive days (Days -3 and -2)
  Arms: BuCy2
Drug: VP-16 — administered as a single infusion on Day -3. The dose is 60 mg/kg and is calculated on actual body weight unless the patient's weight is >/= 150% of IBW, in which case adjusted body weight will be used.
  Other Names: Etoposide (VP-16; Vepesid(R) brand only)
  Arms: VP16/TBI
Radiation: Fractionated Total Body Irradiation (FTBI) — FTBI is performed on day -7 through day -4. The total dose of radiation is 1,320 cGy.
  Arms: VP16/TBI

SUMMARY:
RATIONALE: Giving chemotherapy drugs and total-body irradiation before a donor bone marrow transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

PURPOSE: This phase II trial is studying how well donor bone marrow transplant works in treating patients with hematologic cancers.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the progression free survival (PFS) and overall survival (OS) of patients with low risk myeloid disorders or older allogeneic recipients who are treated with high dose busulfan and cyclophosphamide and allogeneic bone marrow transplantation (BMT).
* Determine the PFS and OS in patients with lymphoid and high risk myeloid disorders who are treated with etoposide, total body irradiation, and allogeneic BMT.
* Evaluate the toxicities of these 2 regimens when combined with cyclosporine and methotrexate as graft versus host disease prophylaxis in these patients.
* Evaluate the PFS and OS of allogeneic BMT in patients with multiple myeloma and chronic lymphocytic leukemia.

OUTLINE:

* Regimen A: Patients with chronic myelogenous leukemia (CP1, AP/CP2) and other myeloproliferative disorders, myelodysplastic disorders, acute myelogenous leukemia (CR1), or multiple myeloma (not eligible to receive total body irradiation due to prior radiation) are treated with high dose busulfan and cyclophosphamide followed by allogeneic bone marrow transplantation (BMT). Patients receive oral busulfan every 6 hours on days -7 to -4 and cyclophosphamide IV over 1 hour on days -3 and -2. Allogeneic bone marrow is infused on day 0.
* Regimen B: Patients with acute myelogenous leukemia (at least CR2, relapsed), acute lymphoid leukemia (ALL), any acute leukemia with CNS involvement, multiple myeloma, or chronic lymphocytic leukemia are treated with total body irradiation and etoposide followed by allogeneic BMT. Patients receive total body irradiation (TBI) on days -7 to -4 for a total of 11 fractions and etoposide IV over 4 hours on day -3. Male patients with ALL receive a testicular boost in 2 fractions on 2 successive days during TBI. Allogeneic bone marrow is infused on day 0.

Patients in both regimens receive cyclosporine and methotrexate as graft versus host disease prophylaxis.

Patients are followed weekly for 3 months and then monthly for 1 year.

PROJECTED ACCRUAL: At least 50 patients with low risk myeloid disease, 50 patients with lymphoid malignancies, and 60 patients with high risk myeloid disease will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of:

  * Acute myelogenous leukemia

    * Complete remission (CR) 1 - ALL except good cytogenetics defined as [(inv16, t(8,21), t(15,17)]
    * CR2
    * Induction failures
    * Relapsed OR
  * Acute lymphocytic leukemia (ALL)

    * CR1 - high risk defined as overt CNS involvement, 1 or more risk factors (age 30 and over, WBC at least 20,000/mm^3, at least 4 weeks to CR1, myeloid phenotype)
    * CR2
    * Induction failures
    * Relapsed OR
  * Chronic myelogenous leukemia

    * Chronic phase (CP) 1
    * Accelerated phase (AP)/CP2 OR
  * Chronic lymphocytic leukemia

    * At diagnosis - RAI stage III/IV or Binet C

      * Must undergo 1 induction regimen
    * Relapsed - any stage

      * Must have received no more than 3 regimens for diagnosis OR
  * Multiple myeloma

    * At diagnosis - stage II/III (primary refractory or sensitive)
    * Relapsed no more than 2 times - sensitive disease
    * Plasma cell leukemia OR
  * Myelodysplasia

    * All subtypes eligible OR
  * Myeloproliferative disorders

    * Poor response to medical therapy OR
    * Cytogenetic abnormalities
* Must have a related donor who is genotypic 6 out of 6 HLA A, B, and DR match

  * Molecular DR matching required

PATIENT CHARACTERISTICS:

Age:

* 15 to 55

Performance status:

* Karnofsky 80-100%

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGOT/SGPT no greater than 3 times upper limit of normal
* PT/PTT normal

Renal:

* Creatinine no greater than 2.0 mg/dL
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* LVEF at least 45% by MUGA scan or echocardiography
* No myocardial infarction within the past 6 months
* No arrhythmias controlled by therapy

Pulmonary:

* FEV_1 at least 50% predicted
* DLCO at least 50% predicted

Other:

* Not pregnant or nursing
* Negative pregnancy test
* No diabetes mellitus or thyroid disease that is not medically controlled
* No psychosocial disorder that would preclude study compliance
* No active serious infections
* HIV negative
* Donor must be HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 1993-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival | 5 years post transplant
  Relapse free survival 5 post transplant deteremiend by the Kaplan-Meier product-limit method.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Field, MD, PhD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida, United States